CLINICAL TRIAL: NCT02787499
Title: Resistance Testing Versus Adherence Support for Management of Patients With Virologic Failure on First-Line Antiretroviral Therapy in Sub-Saharan Africa
Brief Title: Resistance Testing to Improve Management of Virologic Failure in Sub-Saharan Africa
Acronym: REVAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); University of KwaZulu (Other); Emory University (Other); University of Rochester (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mark Siedner, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P000589; R01AI124718 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: HIV; AIDS
Keywords: Drug resistance; Standard of care; sub-saharan africa; antiretroviral therapy; diagnostics; implementation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Follows the 2013 World Health Organization (WHO) HIV treatment guidelines. Study participants will receive adherence support and return for a repeat viral load test in 3 months (or in 1 month for pregnant participants). Treatment failure will be defined by two consecutive viral load measurements greater than 1,000 copies/mL. Participants who meet this criteria will be switched to second-line therapy. Those with a viral load <1,000 copies/mL at repeat testing will be retained on first-line therapy.
- HIV-1 RNA Resistance Testing (Experimental): Participants will receive HIV-1 RNA drug resistance testing at study enrollment. ART treatment regimen decisions will be determined based on the results of resistance testing.
  Interventions: Procedure: HIV-1 RNA Resistance Testing

INTERVENTIONS:
Procedure: HIV-1 RNA Resistance Testing — Perform drug resistance on enrollment to guide management of virologic failure
  Arms: HIV-1 RNA Resistance Testing

SUMMARY:
The study design is an open-label, randomized controlled trial. The study will be conducted at study sites in Uganda and South Africa. The study population will include HIV-infected patients on first-line antiretroviral therapy with a recent viral load >1,000 copies/milliliter (or dried blood spot viral load >1,000 copies/milliliter). Eligible participants will be randomized to the WHO-based standard of care for management of virologic failure or immediate resistance testing to guide ART regimen decisions. The primary outcome of interest will be viral suppression (<200 copies/mL) at 9 months after study enrollment, and will be assessed using an intention to treat analysis, where missing or absent results will be considered failures. Secondary outcomes of interest will be viral suppression below the limit of assay detection, viral suppression on continuation of first-line (non-nucleoside reverse transcriptase inhibitor [NNRTI]-based) therapy, drug resistance at study conclusion, and mortality, among others. The overarching goal of this study is to determine whether addition of routine resistance testing, to guide management of virologic failure and sustain the successful completion of the HIV continuum of care, improves clinical outcomes and reduces costs for patients with virologic failure on first-line therapy in sub-Saharan Africa.

DETAILED DESCRIPTION:
STUDY PROCEDURES FOR PARTICIPANTS RANDOMIZED TO STANDARD OF CARE ARM

A. Visit 1-SOC: Baseline Visit for Standard of Care Participants

At Study Visit 1, participants randomized to the SOC will complete the baseline questionnaire to collect sociodemographic, HIV clinical and treatment history, self-reported ART medication adherence, quality of life, and resource allocation data. Study staff will review participant records to collect data on clinic initiation start date, opportunistic infection history, ART initiation date, ART regimen history, CD4 count and viral load result histories. A single 10cc blood specimen will be drawn for storage for future testing for viral load, resistance testing, and drug therapeutic monitoring. Upon completion of the baseline questionnaire, participants will be referred to clinic counselors who will conduct adherence support counseling as per standard clinical procedures. A follow-up study visit will be scheduled 3 months from the baseline date (or at 1 month for pregnant participants only). Any interim clinical visits that are indicated by the clinic staff will be maintained. The participant will be instructed to continue their current ART regimen until at least the next clinical visit.

B. Visit 2A-SOC: Repeat Viral Load Testing Visit

At Study Visit 2A, participants in the SOC arm will undergo blood collection for viral load testing in keeping with WHO guidelines. An additional tube 10cc tube will be drawn for storage for future analyses. A study questionnaire will be administered to assess self-reported ART medication adherence. No other procedures are scheduled at this visit. Participants will be notified that study staff will contact them as soon as their results are available, to request return to clinic for further management. The participant will be instructed to continue their current ART regimen until at least the next clinical visit. As soon as the viral load result is available, study participants will be contacted and requested to return to clinic for review. If the viral load is indeterminate or not completed for any reason, study staff will request that the participant return for a repeat viral load test.

C. Visit 2B-SOC: Viral Load Testing Results and Therapeutic Management

At Study Visit 2B, study clinicians will review the viral load result. Participants with a viral load ≤ 1,000 copies/mL will continue their first-line (NNRTI-based) ART regimen without change. Participants with a viral load >1,000 copies/mL will change ART regimen to a second-line, protease inhibitor (PI)-based or, if available, integrase inhibitor (II)-based therapy. Clinicians will also be encouraged to change the nucleos(t)ide reverse transcriptase component of the regimen (for example, changing from zidovudine to tenofovir), based on prior exposures, as well as WHO and national guidelines. All regimen decisions will be made by the study clinician, in cooperation with clinic staff at the study sites. In the case of complex management issues, the site principal investigators (Dr. Bosco Bwana in Mbarara and Dr. Yunus Moosa in Durban) will be contacted to offer input. At the conclusion of Visit 2B-SOC, participants in the SOC arm will be scheduled for a final study visit approximately 6 months later. A final visit at 6 months is chosen to allow ample time for drug suppression for participants with detectable viral load at this 3-month visit. Non-study clinical visits for routine clinical care will continue in the interim as determined and scheduled by clinic staff.

D. Visit 3: Outcome Assessment

At Study Visit 3, participants will undergo repeat blood testing for plasma viral load and, if the viral load is detectable, reflex resistance testing will be performed. An additional 10cc tube will be drawn for storage for future testing. A study questionnaire will be administered to assess resource allocation, ART medication adherence, and quality of life. Study staff will review participant records to update interim CD4 count, viral load, and ART regimen data. Results of viral load and resistance testing from this visit will be immediately made available to clinic staff for further patient management. At the conclusion of Visit 3, study procedures will be complete.

E. Missing and Late Appointments

If study participants do not return for study visits, study staff will call them to encourage return to clinic for continuation or completion of procedures. For participants who do not return within 7 days of a scheduled visit and unreachable by phone, a study staff member will attempt to track them at home using a standardized lost-to-follow-up form and procedures developed and used successfully both for program and clinical care in Mbarara for over 10 years. If participants are located, study staff will encourage them to return to clinic to complete procedures and/or conduct the blood draw and questionnaire in in the field if the participant agrees.

STUDY PROCEDURES FOR PARTICIPANTS RANDOMIZED TO RESISTANCE TESTING ARM

A. Visit 1-RT: Baseline Visit for Resistance Testing Participants

At Study Visit 1, participants randomized to the RT will complete the baseline questionnaire to collect sociodemographic, HIV clinical and treatment history, self-reported ART medication adherence, quality of life, and resource allocation data. Study staff will review participant records to collect data on clinic initiation start date, opportunistic infection history, ART initiation date, ART regimen history, CD4 count and viral load result histories. Upon completion of the baseline questionnaire, participants will undergo phlebotomy for resistance testing. Participants will be notified that study staff will contact them as soon as their results are available, to request return to clinic for further management. Upon completion of the study procedures, participants will be referred to clinic counselors who will conduct adherence support counseling as per standard clinical procedures. The participant will be instructed to continue their current ART regimen until at least the next clinical visit. As soon as the resistance test result is available, study participants will be contacted by phone and requested to return to clinic for review.

B. Visit 2-RT: Resistance Testing Results and Therapeutic Management

At Study Visit 2-RT, study clinicians will review the resistance testing result. A study HIV-1 RNA drug resistance interpretation guide will be used to help guide decision-making. Participants without significant drug resistance, as determined by the study clinician in consultation with the resistance interpretation guide will continue their first-line (NNRTI-based) ART regimen without change. Participants with therapeutic drug resistance will change ART regimen to a second-line, protease inhibitor (PI)-based or, if available, integrase inhibitor (II)-based therapy. Clinicians will also be encouraged to change the nucleos(t)ide reverse transcriptase component of the regimen (for example, changing from zidovudine to tenofovir). All regimen decisions will be made by the study clinician, in cooperation with clinic staff at the study sites. In the case of complex management issues, the site principal investigators (Dr. Bosco Bwana in Mbarara and Dr. Yunus Moosa in Durban) will be contacted to offer input. At the conclusion of Visit 2-RT, participants will be scheduled for a final study visit approximately 9 months from the time of enrollment. A final visit 9 months later is chosen to match the approximate 9-month study duration for participants in the SOC arm. Non-study clinical visits for routine clinical care will continue in the interim as determined and scheduled by clinic staff.

C. Visit 3: Outcome Assessment

At Study Visit 3, participants will undergo repeat blood testing for plasma viral load and, if the viral load is detectable, reflex resistance testing will be performed. An additional 10cc tube will be drawn for storage for future testing for viral load, resistance testing, and drug therapeutic monitoring. A study questionnaire will be administered to assess resource allocation and quality of life. Study staff will review participant records to update interim CD4 count, viral load, and ART regimen data. Results of viral load and resistance testing from this visit will be immediately made available to clinic staff for further patient management. At the conclusion of Visit 3, study procedures will be complete.

ELIGIBILITY:
Inclusion Criteria:

* In care at a public HIV clinic within a PEPFAR-focus sub-Saharan African country (South Africa or Uganda) and living within 100 kilometers of the clinic
* Age ≥ 18 years at the time of enrollment
* Currently prescribed first-line (non-nucleoside reverse transcriptase inhibitor [NNRTI]-based) ART for at least 5 months. Switches within first line regimens, including NNRTI and nucleos(t)ide backbone changes are allowed.
* Detectable plasma viral load > 1,000 copies/mL or dried blood spot viral load > 1,000 copies/mL within 90 days of enrollment

Exclusion Criteria:

* Known prior drug resistance
* Prior exposure to PI-based ART
* Current clinical indication to start PI-based ART
* Not planning to remain in the clinic catchment area for the next nine months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mwebesa Bwana, MBChB MPH, Principal Investigator — Mbarara University of Science and Technology; Yunus Moosa, MBChB PhD, Principal Investigator — University of KwaZulu
Locations (2):
- University of Kwa-Zulu Natal, Durban, South Africa
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will be made public and accessible through request after completion of primary analysis.
Time Frame: Data will become publicly available after study completion.
Access Criteria: Publicly available
URL: https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/SKUUOP

REFERENCES:
- [Background] Rautenberg TA, George G, Bwana MB, Moosa MS, Pillay S, McCluskey SM, Aturinda I, Ard K, Muyindike W, Moodley P, Brijkumar J, Johnson BA, Gandhi RT, Sunpath H, Marconi VC, Siedner MJ. Comparative analyses of published cost effectiveness models highlight critical considerations which are useful to inform development of new models. J Med Econ. 2020 Mar;23(3):221-227. doi: 10.1080/13696998.2019.1705314. Epub 2020 Jan 11. PMID 31835974
- [Background] Siedner MJ, Bwana MB, Moosa MS, Paul M, Pillay S, McCluskey S, Aturinda I, Ard K, Muyindike W, Moodley P, Brijkumar J, Rautenberg T, George G, Johnson B, Gandhi RT, Sunpath H, Marconi VC. The REVAMP trial to evaluate HIV resistance testing in sub-Saharan Africa: a case study in clinical trial design in resource limited settings to optimize effectiveness and cost effectiveness estimates. HIV Clin Trials. 2017 Jul;18(4):149-155. doi: 10.1080/15284336.2017.1349028. Epub 2017 Jul 18. PMID 28720039
- [Result] Siedner MJ, Moosa MS, McCluskey S, Gilbert RF, Pillay S, Aturinda I, Ard K, Muyindike W, Musinguzi N, Masette G, Pillay M, Moodley P, Brijkumar J, Rautenberg T, George G, Gandhi RT, Johnson BA, Sunpath H, Bwana MB, Marconi VC. Resistance Testing for Management of HIV Virologic Failure in Sub-Saharan Africa : An Unblinded Randomized Controlled Trial. Ann Intern Med. 2021 Dec;174(12):1683-1692. doi: 10.7326/M21-2229. Epub 2021 Oct 26. PMID 34698502
- [Result] Reynolds Z, McCluskey SM, Moosa MYS, Gilbert RF, Pillay S, Aturinda I, Ard KL, Muyindike W, Musinguzi N, Masette G, Moodley P, Brijkumar J, Rautenberg T, George G, Johnson BA, Gandhi RT, Sunpath H, Marconi VC, Bwana MB, Siedner MJ. Who's slipping through the cracks? A comprehensive individual, clinical and health system characterization of people with virological failure on first-line HIV treatment in Uganda and South Africa. HIV Med. 2022 May;23(5):474-484. doi: 10.1111/hiv.13203. Epub 2021 Nov 9. PMID 34755438
- [Derived] Rautenberg TA, Ng SK, George G, Moosa MS, McCluskey SM, Gilbert RF, Pillay S, Aturinda I, Ard KL, Muyindike WR, Musinguzi N, Masette G, Pillay M, Moodley P, Brijkumar J, Gandhi RT, Johnson B, Sunpath H, Bwana MB, Marconi VC, Siedner MJ. Determinants of health-related quality of life in people with Human Immunodeficiency Virus, failing first-line treatment in Africa. Health Qual Life Outcomes. 2023 Aug 21;21(1):94. doi: 10.1186/s12955-023-02179-x. PMID 37605150
- See also: De-identified Participant Data Set — https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/SKUUOP
- Available data/document: Individual Participant Data Set — https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/SKUUOP — Publicly available, de-identified datasets are available on the Harvard Dataverse Platform.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Started | 423 | 417
Completed | 423 | 417
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing | Total
Number analyzed (Participants) | 423 | 417 | 840
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 415 | 412 | 827
  >=65 years | 4 | 3 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [31 to 45] | 37 [30 to 44] | 37 [31 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 209 | 430
  Male | 202 | 208 | 410
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 423 | 417 | 840
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 210 | 210 | 420
  South Africa | 213 | 207 | 420
Median Antiretroviral therapy (ART) duration [Median (Inter-Quartile Range); unit: years] | 3.5 [1.1 to 6.5] | 3.0 [1.1 to 6.4] | 3.2 [1.1 to 6.4]
Country [Count of Participants; unit: Participants]
  Uganda | 210 | 210 | 420
  South Africa | 213 | 207 | 420
Pregnancy [Count of Participants; unit: Participants]
  Pregnant at enrollment | 7 | 6 | 13
  Not pregnant at enrollment | 416 | 411 | 827
Median CD4 count [Median (Inter-Quartile Range); unit: x 10^9 cells/L] | 0.303 [0.132 to 0.475] | 0.259 [0.112 to 0.434] | 0.281 [0.121 to 0.457]
ART regimen [Count of Participants; unit: Participants]
  TDF-3(F)TC-EFV | 311 | 295 | 606
  AZT-3TC-NVP | 60 | 58 | 118
  Other | 52 | 64 | 116
Self-reported treatment adherence at enrollment [Count of Participants; unit: Participants]
  <100% in prior 30 d | 297 | 295 | 592
  100% in prior 30 d | 126 | 122 | 248

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Patients Achieving Virologic Resuppression
Description: Number and percentage of participants achieving virologic suppression. Virologic resuppression defined as viral load < 200 copies/mL
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
Participants | 256 | 263

2. Secondary Outcome: Number and Percentage of Patients With an Undetectable Viral Load (Below Limit of Detection) at Study Conclusion
Description: Number and percentage of patients with an undetectable viral load (below limit of detection) at study conclusion. Viral load < 200 copies/mL
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
Participants | 193 | 202

3. Secondary Outcome: Number and Percentage of Patients With an Undetectable Viral Load on First-line (NNRTI-based) Therapy at Study Conclusion
Description: The number and percentage of patients with an undetectable viral load on first-line (NNRTI-based) therapy at study conclusion. Viral load < 200 copies/mL
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
Participants | 81 | 62

4. Secondary Outcome: Number and Percentage of Patients With International AIDS Society-defined Drug Resistance Mutations to Their Current Regimen.
Description: Proportion of patients with International AIDS Society-defined drug resistance mutations to their current regimen. As part of this analysis, we will also evaluate for minority drug resistance
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 103 | 82
Participants | 25 | 34

5. Secondary Outcome: Total Patient Care Costs, Including Diagnostic Testing and ART Costs for the Study Duration
Description: Total patient care costs, including diagnostic testing and ART costs for the study duration. These data are reported as median cost and IQR per person by arm.
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
dollars | 227 [124 to 416] | 400 [304 to 579]

6. Secondary Outcome: Number and Percentage of Patients Retained in HIV Clinical Care at Study Completion
Description: The number and percentage of patients retained in HIV clinical care at study completion
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
Participants | 403 | 394

7. Secondary Outcome: Number and Percentage of Participants Survived Through 9-month Study Period
Description: Odds of 9-month survival. Number and percentage of participants who survived through the 9-month (then 15-month) study period.
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 423 | 417
Participants | 415 | 403

8. Secondary Outcome: Change in Health-related Quality of Life From Baseline to 9 Months
Description: Change in health-related quality of life from baseline to 9 months. The scale used is Health-related Quality of Life (HRQoL), where the minimum score is 0 = 'death' and the maximum is 1 = 'perfect' health. We are reporting mean change in HRQoL, so a larger positive value indicates a larger improvement of HRQoL. Two time points used in the calculation were the HRQoL score at the baseline visit and at the final visit at 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic).
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Population: This analysis was completed for participants with complete utility data at visit 3 (at 9 months or 15 months due to the pandemic). There was missing HRQoL data for 24 participants in the Standard of Care arm and 19 participants in the Resistance Testing arm at visit 3. Therefore, the numbers of participants for this outcome are different from other outcome measures.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
Number analyzed (Participants) | 399 | 398
score on a scale | 0.064 [0.042 to 0.086] | 0.078 [0.053 to 0.102]

ADVERSE EVENTS:
Time Frame: 9 months (end point extended up to 15 months for participants affected by the COVID-19 epidemic)
Arm/Group | Standard of Care | HIV-1 RNA Resistance Testing
All-Cause Mortality (participants affected / at risk) | 8/423 | 14/417
Serious Adverse Events (participants affected / at risk) | 0/423 | 0/417
Other Adverse Events (participants affected / at risk) | 0/423 | 0/417

LIMITATIONS AND CAVEATS:
The study underwent a single major protocol change in 2020, when the study window was extended for participants who were actively enrolled in the trial but unable to return to the clinic for their outcome assessment while COVID-19 transportation restrictions were imposed in both countries (24 March 2020 in Uganda and 27 March 2020 in South Africa.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT02787499/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT02787499/ICF_001.pdf